CLINICAL TRIAL: NCT01597921
Title: Phase II, Double Blinded, Randomized Study of R1 and R2 (Waterjel) Verses Aloe Vera Jell for the Prevention and Treatment of Radiation Induced Dermatitis in Breast Cancer Patients
Brief Title: A DB Randomized Study of R1 and R2 WaterJel / AloeVera Jell in Prevention of Radiation Dermatitis in Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: The study was stopped due to unbalanced side effects
Sponsor: Water-Jel (Industry)
Responsible Party: Principal Investigator, Dr Merav Ben-David, Dr, Water-Jel
Other Study IDs: 23267384
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer; Radiation Dermatitis; Erythema
Keywords: Breast conserving surgery; Radiation dermatitis
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis; Erythema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patient receiving RT: Total dose:2Gy/Fx

SUMMARY:
The purpose of this study is to evaluate the effects of topical R1 and R2 for prophylaxis of acute radiation dermatitis in patients with breast cancer receiving radiotherapy.

DETAILED DESCRIPTION:
All women will be given two types of Jell. One should be applied immediately after radiation and the second one, 3 times every day. All women will complete detailed questionnaire every two weeks and will be evaluated by the treating team at the same time.All women will be evaluated two weeks after end of radiation period.

ELIGIBILITY:
Inclusion Criteria:

1. Woman with histologically confirmed breast cancer who underwent lumpectomy and requires adjuvant radiation therapy with 2 Gy/fx to a total dose of 50 Gy.
2. Women who received neoadjuvant or adjuvant chemotherapy are eligible for the study. Three weeks is the minimal interval between chemotherapy and start of radiation therapy.
3. Patient able to understand the study designed and cooperate with instructions of use.
4. Patient able to sign informed consent

Exclusion Criteria:

1. Woman with lactose allergy (lactose intolerance are eligible)
2. Woman with known connective tissue disorder
3. Woman with uncontrolled diabetes
4. Patients receiving radiation protocol with 2.64 Gy/fx or 1.8 Gy/fx
5. Woman who is unable to sign an informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 75
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Merav Ben David, Principal Investigator — La Sheba Hospital
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel